CLINICAL TRIAL: NCT00104741
Title: Multicentre Randomized Trial Assessing the Efficacy of a Short Neoadjuvant and Concomitant Hormone Therapy to an Exclusive Curative Cornformational Radiotherapy of Locolized Prostate Cancer With Intermediate Prognosis
Brief Title: Triptorelin, Flutamide, and External-Beam Radiation Therapy or External-Beam Radiation Therapy Alone in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/0207; FRE-FNCLCC-GETUG-14/0207; EU-20503
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Triptorelin Pamoate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiotherapy alone (Active Comparator)
  Interventions: Radiation: radiation therapy
- Radiotherapy + androgene deprivation (Experimental)
  Interventions: Drug: flutamide; Drug: triptorelin; Radiation: radiation therapy

INTERVENTIONS:
Drug: flutamide
  Arms: Radiotherapy + androgene deprivation
Drug: triptorelin
  Arms: Radiotherapy + androgene deprivation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as triptorelin and flutamide, may stop the adrenal glands from making androgens. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving triptorelin and flutamide together with radiation therapy may be an effective treatment for prostate cancer. It is not yet known whether giving triptorelin and flutamide together with external-beam radiation therapy is more effective than external-beam radiation therapy alone in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying triptorelin, flutamide, and external-beam radiation therapy to see how well they work compared to external-beam radiation therapy alone in treating patients with stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the impact of neoadjuvant androgen blockade therapy comprising triptorelin and flutamide followed by conformal external beam radiotherapy and continued androgen blockage therapy vs conformal external beam radiotherapy alone in patients with stage II or III prostate cancer.
* Compare the survival rate, in terms of 5-year clinical or biological remission, in patients treated with these regimens.
* Compare overall survival in patients treated with these regimens.
* Compare acute and late toxicity of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.
* Determine the value and time-delay to obtain prostate-specific antigen nadir in patients treated with external beam radiotherapy alone.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo conformal external beam radiotherapy.
* Arm II: Patients receive androgen blockade therapy comprising triptorelin subcutaneously every 4 weeks and oral flutamide once daily. Androgen blockade therapy continues for a total of 4 months. Two months after initiation of androgen blockade therapy, patients undergo conformal external beam radiotherapy.

Quality of life is assessed.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer, meeting the following clinical staging criteria:

  * Stage T1b-T1c AND prostate specific antigen (PSA) ≥ 10 ng/mL OR Stage T1b-T1c AND Gleason score ≥ 7 OR Stage T2a-T3a
  * No lymph node invasion (N0 or N-)

    * Patients with ≥ 10% risk by the Partin table must undergo curage
  * No metastatic disease (M0) by thoracic radiography and bone scan
* PSA < 30 ng/mL
* No history of invasive cancer

PATIENT CHARACTERISTICS:

Age

* Under 75

Performance status

* ECOG 0-1

Life expectancy

* At least 10 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior hormonal therapy

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* No prior radical prostatectomy
* No prior castration

Ages: 0 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2003-09-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10-15 (Actual)

PRIMARY OUTCOMES:
Impact of complete androgen blockade for 4 months
Survival, in terms of clinical or biological remission, at 5 years
Overall survival
Acute and late toxicity
Quality of life
Value and time-delay to obtain prostate-specific antigen nadir (for patients undergoing external beam radiotherapy alone)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard M. Dubray, MD, PhD, Study Chair — Centre Henri Becquerel
Locations (31):
- France (31):
  - Clinique De Rochebelle, Alès
  - Institut Sainte Catherine, Avignon
  - Hopital Louis Pasteur, Colmar
  - Hopitaux Civils de Colmar, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Intercommunal De Creteil, Créteil
  - Hopital Jean Monnet, Épinal
  - Centre Hospitalier Intercommunal des Alpes du Sud, Gap
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Hospitalier, Mulhouse
  - Centre Regional Rene Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Clinique De Valdegour, Nîmes
  - Hopital d'Instruction des Armees du Val de Grace, Paris
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Campillo-Gimenez B, Buscail C, Zekri O, Laguerre B, Le Prise E, De Crevoisier R, Cuggia M. Improving the pre-screening of eligible patients in order to increase enrollment in cancer clinical trials. Trials. 2015 Jan 16;16:15. doi: 10.1186/s13063-014-0535-7. PMID 25592642